CLINICAL TRIAL: NCT05318846
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Phase IIa Clinical Trial to Evaluate the Efficacy and Safety of HRS4800 Tablets for Postoperative Analgesia After Impacted Teeth Removal Surgery
Brief Title: A Study to Evaluate the Efficacy and Safety of HRS4800 Tablets for Postoperative Analgesia After Impacted Teeth Removal Surgery.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HRS4800-201
Record Dates: First submitted 2022-03-04; First posted 2022-04-08 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-03

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: A multicenter, randomized, double-blind, placebo-controlled, phase IIa clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group A (Experimental)
  Interventions: Drug: HRS4800 tablets
- Treatment group B (Placebo Comparator)
  Interventions: Drug: Placebo tablets

INTERVENTIONS:
Drug: HRS4800 tablets — Dosing frequency: single dose; Route of administration: oral
  Arms: Treatment group A
Drug: Placebo tablets — Dosing frequency: single dose; Route of administration: oral
  Arms: Treatment group B

SUMMARY:
The study is being conducted to evaluate the efficacy and safety of HRS4800 tablets for postoperative analgesia after impacted teeth removal surgery.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 65 years old.
2. Scheduled to remove the impacted tooth.
3. Any NRS score ≥5 within 4 hours after the surgery.
4. Willing to comply with the study procedures and requirements.
5. Willing and able to provide written informed consent for this study.

Exclusion Criteria:

1. Subjects who had used other drugs that affect the analgesic effect.
2. Subjects who have infection or other complications on the planned oral surgical site.
3. Subjects with uncontrolled hypertension or hypotension.
4. Subjects with severe cardiovascular and cerebrovascular diseases.
5. Subjects with severe gastrointestinal disease.
6. Subjects with a history of drug or alcohol abuse.
7. Subjects with significant abnormal electrocardiogram.
8. Subjects with significant abnormal laboratory value.
9. Subject who were allergic to the study drug and ingredients.
10. Pregnancy, lactation or having recent pregnant plan.
11. Subjects who participated in other clinical research study 30 days before entering this study.
12. Other conditions unsuitable for participation in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2022-01-14 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-03-22 (Actual)

PRIMARY OUTCOMES:
the Sum of Pain Intensity Differences (SPID) using numerical rating scale (NRS, ranging from 0-10, the larger the number, the more severe the pain) 0-8 hours after drug administration | 0-8 hours after drug administration

SECONDARY OUTCOMES:
the Differences of Pain Intensity (PID) form each evaluating timepoint to baseline using numerical rating scale (NRS, ranging from 0-10, the larger the number, the more severe the pain) after drug administration | 0-12 hours after drug administration
the Sum of Pain Intensity Differences (SPID) using numerical rating scale (NRS, ranging from 0-10, the larger the number, the more severe the pain) 0-4 hours after drug administration | 0-4 hours after drug administration
the Sum of Pain Intensity Differences (SPID) using numerical rating scale (NRS, ranging from 0-10, the larger the number, the more severe the pain) 0-12 hours after drug administrationadministration | 0-12 hours after drug administration
Pain relief degree at each evaluating timepoint using pain relief scale (PAR, ranging from 0-4, the larger the number, the more obvious the pain relief) after drug administration | 0-12 hours after drug administration
Sum of pain relief degree within 4 hours using pain relief scale (PAR, ranging from 0-4, the larger the number, the more obvious the pain relief) after drug administration (SPAR) | 0-4 hours after drug administration
Sum of pain relief degree within 8 hours using pain relief scale (PAR, ranging from 0-4, the larger the number, the more obvious the pain relief) after drug administration (SPAR) | 0-8 hours after drug administration
Sum of pain relief degree within 12 hours using pain relief scale (PAR, ranging from 0-4, the larger the number, the more obvious the pain relief) after drug administration (SPAR) | 0-12 hours after drug administration
Proportion of subjects who reaches a 50% reduction in pain intensity from baseline using numerical rating scale (NRS, ranging from 0-10, the larger the number, the more severe the pain) at each evaluating timepoint | 0-12 hours after drug administration
Time from drug administration to the first NRS score≤3 | 0-12 hours after drug administration
Time from drug administration to the first use of rescue medication | 0-12 hours after drug administration
Proportion of subjects who receive rescue therapy during the treatment period | 0-12 hours after drug administration
Subject's overall satisfaction score of the study medication using subject satisfaction scale (ranging from 0-10, the larger the number, the higher the satisfaction) | 12 hours after drug administration

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Stomatology Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided